CLINICAL TRIAL: NCT04883398
Title: Neural and Cognitive Mechanisms of Attention and Memory Deficits in Cancer Survivors
Brief Title: A Study of Attention and Memory Processes in Breast Cancer Survivors
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Baruch College City University of New York (Other)
Responsible Party: Sponsor
Other Study IDs: 21-161
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Survivors
Keywords: Neural and Cognitive Mechanisms; Memory Deficits; 21-161
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer survivors: Breast cancer survivors ages 50-70 with AJCC stages 0-3 breast cancer who are at least 1 year post-treatment (including surgery, radiation, and chemotherapy, with or without current endocrine therapy)
- Healthy controls: Healthy controls ages 50-70 with no history of cancer.

SUMMARY:
The purpose of this study is to observe the attention and memory processes in breast cancer survivors. Both cancer survivors and healthy volunteers (who are the same age as the cancer survivors) will participate in this study so we can compare the results of testing on each group of participants.

ELIGIBILITY:
Inclusion Criteria:

For All Paricipants:

* As per medical record or self-report, female
* As per medical record or self-report, age 50-70
* Score of < 11 on the Blessed Orientation-Memory-Concentration Test (BOMC)
* English fluent (as per self reported fluency of "well" or "very well", and having a reasonable comprehension of the study conversation in the opinion of the research staff/preference of English language for healthcare)**
* As per medical record or self-report, if currently taking psychoactive medications (excluding gabapentin and including but not limited to antidepressants and anxiolytics) on a daily basis, dose must have been stable at least two months prior to enrollment

For Survivors:

* As per medical record or self-report, AJCC stages 0-3 breast cancer
* As per medical record or self-report, at least 1-year post-treatment for breast cancer (including surgery, and chemotherapy, with or without radiation
* As per medical record or self-report, current endocrine therapy

For Healthy Controls:

* As per self-report, if currently taking psychoactive medications (including but not limited to antidepressants and anxiolytics), dose must have been stable at least two months prior to enrollment.
* As per self report, no history of cancer except non-melanoma/basal cell skin cancer/squamous cell skin carcinoma

Exclusion Criteria:

For All Participants:

* As per medical record or self-report, diagnosis of neurodegenerative disorder that affects cognitive function (e.g. Alzheimer's disease, Parkinson's disease, Multiple Sclerosis, Dementia, Seizure Disorders, etc.)
* As per medical record or self report, history of stroke or head injury resulting in a structural lesion on neuropsych imaging, persistent cognitive difficulties impacting work or daily life, or required cognitive rehabilitation
* As per medical record or self report, a diagnosis of a Schizophrenia Spectrum Disorder, substance use disorder, Bipolar Disorder or Schizotypal personality disorder. Schizophrenia Spectrum Disorders include Schizophrenia, Schizophreniform disorder, Schizoaffective disorder, Delusional disorder, Brief psychotic disorder, and Attenuated Psychotic Disorder
* As per medical record or self-report, visual or auditory impairment that would preclude ability to complete the assessments (e.g. history of significant macular degeneration or being unable to correct hearing with hearing aides)
* As per medical record or self-report, use of methotrexate (Amethopterin, Rhematrex, Trexall) or rituximab (Rituxin) for rheumatoid arthritis, psoriasis or Crohn's disease, or cyclophosphamide (Cytoxan, Neosar) for Lupus
* As per medical record or self-report, participation in a conflicting research study (i.e. another neurocognitive study utilizing HVLT and BVMT tasks.)

For Survivors only:

* As per medical record or self-report, history of another type of cancer or prior breast cancer diagnosis except non-melanoma/basal cell skin cancer/squamous cell skin carcinoma
* As per medical record or self-report, disease recurrence.

For Healthy Controls only:

* As per medical record or self-report, history of treatment using radiation, chemotherapy, and/or Tamoxifen or Aromatase-inhibitors

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Survivors will be recruited in Breast Medicine Service clinics at the Breast and Imaging Center
Study Population: Breast cancer survivors and Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
test early attentional deficits | baseline
  Using EEG measures of brain activity during a cognitive-experimental long-term memory task to evaluate the mechanisms underlying attention, initial learning, retrieval, and metamemory performance. P3 amplitude as measured by EEG at the Pz electrode.
abnormal event-related potential (ERP) during initial learning | baseline
  During passive tasks (such as a paired-click paradigm)The proposed paradigm is adapted from previous work using EEG to measure the relationship between attention, learning, and subsequent performance on a verbal long-term memory task in healthy adults41. Relative to standard neuropsychological measures, this technique provides a more finely grained approach to investigating the effect of attentional mechanisms on subcomponents of initial learning and retrieval processes in long-term memory.

CONTACTS AND LOCATIONS:
Overall Officials: James Root, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

DOCUMENTS (1):
  • Informed Consent Form (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT04883398/ICF_000.pdf